CLINICAL TRIAL: NCT02214940
Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Multiple, Rising Oral Doses of 2.5 mg, 5 mg, 7.5 mg, and 10 mg BI 11634 Oral Solution Administered t.i.d. for 5 Days to Healthy Male Volunteers; Randomised, Doubleblind, Placebo-controlled at Each Dose Level
Brief Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Multiple, Rising Oral Doses of BI 11634 Oral Solution in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1234.2
Record Dates: First submitted 2014-08-12; First posted 2014-08-13 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
MeSH Terms: interventions — N-(1-(5-chloro-1H-benzimidazol-2-yl)-2-methoxyethyl)-3-methyl-4-(3-oxo-4-morpholinyl)benzamide

ARMS (2):
- BI 11634 (Experimental): multiple rising dose
  Interventions: Drug: BI 11634
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 11634
  Arms: BI 11634
Drug: Placebo
  Arms: Placebo

SUMMARY:
First evaluation of safety, tolerability, pharmacokinetics, and the pharmacodynamic effect of BI 11634 on coagulation parameters after multiple-dose administration (no primary endpoint in a statistical sense defined)

ELIGIBILITY:
Inclusion Criteria:

* Healthy Caucasian males according to the following criteria: Based upon a complete medical history, including the physical examination, vital signs (blood pressure, pulse rate), 12-lead ECG, clinical laboratory tests
* Age ≥18 and ≤50 years
* Haemoglobin within the normal ranges
* Body Mass Index (BMI) ≥18.5 and BMI ≤29.9 kg/m2
* Signed and dated written informed consent prior to admission to the study in accordance with Good clinical practice (GCP) and the local legislation

Exclusion Criteria:

* Relevant gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Relevant surgery of gastrointestinal tract
* History of any bleeding disorder or acute and chronic blood coagulation defect, for the subject itself or any person of his family as far as known
* History of gastric ulcera and cholecystectomy
* Occult blood in feces
* Relevant diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Relevant chronic or acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (>24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
* Use of acetylsalicylic acid or any other non-steroidal anti-inflammatory drugs (NSAID) within 2 weeks of study start until the end of study
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Smoker (>10 cigarettes or >3 cigars or >3 pipes/day)
* Inability to refrain from smoking on trial days as judged by the investigator
* Alcohol abuse (more than 40 g/day)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Vulnerable subjects (e.g. persons kept in detention)
* The subject is not able to understand and comply with protocol requirements, instructions and protocol-stated restrictions
* Subjects with a history within the past six weeks of closed-head or torso trauma or deceleration injury such as an automobile accident or fall from a significant height
* Inability to comply with dietary regimen of the study centre
* Inability to understand the protocol requirements, instructions and study-related restrictions; the nature, scope and possible consequences of the study
* Subjects (including those who have had a vasectomy) who do not agree to use two methods of contraception, including barrier contraception (latex condoms with spermicide plus intrauterine device) when engaging in sexual activity with women of child bearing potential during the study and for 60 days after completion of the study

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2007-06; Primary Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events | up to 10 days after last drug administration
Number of subjects with clinically significant findings in vital signs (blood pressure, pulse rate) | up to 10 days after last drug administration
Number of subjects with clinically significant findings in ECG | up to 10 days after last drug administration
Number of subjects with clinically significant findings laboratory tests | up to 10 days after last drug administration
Assessment of tolerability by investigator on a 4-point scale | up to 10 days after last drug administration

SECONDARY OUTCOMES:
Cmax (maximum measured concentration of analyte in plasma) | up to 144 hours after first drug administration
tmax (time from dosing to maximum measured concentration) | up to 144 hours after first drug administration
AUCτ,n (area under the concentration-time curve of analyte in plasma over a uniform dosing interval τ after administration of the n-th dose) | up to 144 hours after first drug administration
Aet1-t2 (amount of analyte eliminated in urine from the time point t1 to time point t2) | up to 144 hours after first drug administration
fet1-t2 (fraction of analyte eliminated in urine from time point t1 to time point t2) | up to 144 hours after first drug administration
CLR,t1-t2 (renal clearance of analyte from the time point t1 until the time point t2) | up to 144 hours after first drug administration
Cmin,ss (minimum measured concentration of analyte in plasma at steady state over a uniform dosing interval τ) | up to 144 hours after first drug administration
Cpre,ss (predose concentration of analyte in plasma at steady state immediately before administration of the next dose) | up to 144 hours after first drug administration
λz,ss (terminal rate constant in plasma at steady state) | up to 144 hours after first drug administration
t1/2,ss (terminal half-life of analyte in plasma at steady state) | up to 144 hours after first drug administration
MRTpo,ss (mean residence time of analyte in the body after multiple oral administrations at steady state) | up to 144 hours after first drug administration
CL/F,ss (apparent clearance of analyte in the plasma at steady state following extravascular multiple dose administration) | up to 144 hours after first drug administration
Vz/F,ss (apparent volume of distribution during the terminal phase λz at steady state following extravascular administration) | up to 144 hours after first drug administration
PTF (peak-trough fluctuation) | up to 144 hours after first drug administration
Cavg (average concentration of analyte in plasma at steady state) | up to 144 hours after first drug administration
RA,Cmax (Accumulation ratio of analyte in plasma based on Cmax) | up to 144 hours after first drug administration
RA,AUC (Accumulation ratio of analyte in plasma based on AUC) | up to 144 hours after first drug administration
Cpre,N (predose concentration of analyte in plasma immediately before administration of the Nth dose after N-1 doses were administered ) | up to 144 hours after first drug administration
Activated partial thromboplastin time (aPTT) ratios between groups | up to 144 hours after first drug administration
Maximum aPTT prolongation | up to 144 hours after first drug administration
Maximum international normalized ratio (INR) | up to 144 hours after first drug administration
% inhibition of endogenous Factor Xa | up to 144 hours after first drug administration
  by Russel's Viper Venom test (RVV)
Maximum prolongation of blood coagulation time | up to 144 hours after first drug administration
  by HepTest® (Haemachem Inc.)
Percent inhibition of FXa | up to 144 hours after first drug administration
  by COAMATIC© Heparin test (Chromogenix)
Percent inhibition of thrombin generation by BI 11634 | up to 144 hours after first drug administration
Percent peak inhibition of thrombin generation | up to 144 hours after first drug administration
Time to maximum inhibition of thrombin generation BI 11634 | up to 144 hours after first drug administration
Percent prolongation of lag time | up to 144 hours after first drug administration